CLINICAL TRIAL: NCT05741203
Title: Sviluppo di un Sistema di Supporto Alle Decisioni Tramite Software Multiomico Basato su Modelli Preclinici e Dati Point-of-care Clinici e Ecografici Polmonari Per la Gestione Personalizzata Dei Bambini Con Polmonite Acquisita in comunità
Brief Title: Lung Ultrasound in Pediatric CAP
Acronym: ULTRASONIC-CAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 5474
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with LRTI
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — lung ultrasound

SUMMARY:
Community-acquired Pneumonia (CAP) represents the single largest cause of death and morbidity in children worldwide (1). Respiratory viruses are the most common cause of CAP in preschool children, followed by bacteria. The atypical bacteria Mycoplasma pneumoniae and Chlamydia pneumoniae are common causes of pneumonia in children >5 years. The identification of the causal agent is pivotal, especially in children who require hospital admission, as it guides the choice of appropriate treatment. However, the microbial diagnosis of CAP in children is not easy to establish without invasive procedures, and chest X-Ray has failed to identify the aetiology of CAP. Clinical features of bacterial pneumonia, atypical bacterial pneumonia or viral pneumonia frequently overlap and cannot be used reliably to distinguish between the various aetiologies, as well as blood tests like white blood cell, C-reactive protein, including the more recently introduced serum procalcitonin (85% sensitivity and 45% specificity in identifying children without typical bacterial CAP. As a consequence, children with CAP usually receive unnecessary empirical antibiotics, contributing to the spread of antibiotic resistance or to side effects. Therefore, new methods, possibly fast, non- invasive and easily accessible in the outpatient settings (point-of-care) to optimize and personalize the management of children with suspected CAP are urgently needed

Specific aim 1 To perform a clinical prospective study aimed to evaluate clinical, laboratory, microbiolical and outcomes data and to define LUS patterns (ultrasonomic) in children with CAP of different aetiologies: (viral, bacterial and atypical CAP) in different italian regions (Lazio, Puglia).

Specific Aim 2 Development and validation of multi-factorial prediction models for the personalized diagnosis and management of paediatric CAP and building of a Decision Support System (DSS) based on validated prediction models that will be build based on the collection of "ultrasonomic", clinical, laboratory, treatments, outcomes and microbiological data collected from all partners. In particular, we will: i) develop, validate, and improve prediction models for the prediction of aetiology, outcome and treatment response; ii) take advantage of prediction models to better inform patients/caregivers on the risks and benefits of the proposed treatments; iii) use the outcome of the prediction models to individualize the management

ELIGIBILITY:
Inclusion Criteria:

* Bambini con diagnosi clinica di infezione delle basse vie respiratorie acuta (ALRTI) (basata su anamnesi, esame clinico, esami del sangue (se eseguiti) e CXR (se eseguiti) sottoposti a LUS entro sei ore dalla prima valutazione clinica

Exclusion Criteria:

* Pazienti con patologie preesistenti, tra cui anomalie del tratto respiratorio, immunodeficienza, paralisi cerebrale, malattie neuromuscolari, cardiopatie congenite e tumori maligni

Ages: 6 Months to 17 Years | Sex: All
Age Groups: Child
Study Population: Bambini con diagnosi clinica di infezione delle basse vie respiratorie acuta (ALRTI) (basata su anamnesi, esame clinico, esami del sangue (se eseguiti) e CXR (se eseguiti) sottoposti a LUS entro sei ore dalla prima valutazione clinica
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pneumonia aetiology | 2 years
  definition of characteristics predictive of viral vs bacterial pneumonia

IPD SHARING:
Plan to Share IPD: No